CLINICAL TRIAL: NCT04006132
Title: Evaluation of the Benefits of Bilateral Fitting in Bone-anchored Hearing System Users
Brief Title: Evaluation of the Benefits of Bilateral Fitting in BAHS Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C71
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Bilateral Hearing Loss
Keywords: Bone anchored hearing systems; BAHS; Bilateral benefit; Ponto 3 SuperPower; Minimum Audible Angle; Auditory working memory
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Masking Description: The participants are blinded to the tested condition (unilateral vs bilateral)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ponto 3 SuperPower sound processor (Experimental): All patients will be fitted with two bone-anchored sound processors (Ponto 3 SuperPower), unilaterally and bilaterally.
  Interventions: Device: Fitting of Ponto 3 SuperPower

INTERVENTIONS:
Device: Fitting of Ponto 3 SuperPower — Bone-anchored hearing systems (BAHS) use the body's natural ability to transfer sound through bone conduction. The sound processor picks up sound and converts it into vibrations that are transferred through the skull bone to the inner ear (cochlea). Thus, for patients with conductive or mixed hearing losses, patients with lasting hearing loss following a middle ear disease or malformations (such as microtia), the vibrations are bypassing the conductive problem in the ear canal or middle ear. The intervention in this study is audiologically fitting two bone-anchored sound processors (Ponto 3 SuperPower) to patients that are already bilaterally implanted with abutments.

SUMMARY:
The purpose of this study is to evaluate the benefit of bilateral implantation with bone-anchored hearing systems (BAHS), in terms of sound localization abilities, as well as auditory working memory. The hypothesis is that the use of two BAHS (bilateral condition) will not only improve localization abilities, but it will also increase the ability to retain words in working memory, compared to performance with only one BAHS (unilateral condition).

DETAILED DESCRIPTION:
The patients included in this study are adult patients with a bilateral conductive or mixed hearing loss, that are already bilaterally implanted with two percutaneous bone-anchored devices (BAHS). The study consists of two visits. At visit 1, the patients are fitted unilaterally and bilaterally with the investigational device (Ponto 3 SuperPower). After fitting, the patients perform a test of spatial resolution (minimum audible angle, visit 1) and an auditory working memory test (visit 2). These two outcome measures are conducted in the laboratory using the Ponto 3 SuperPower unilaterally and bilaterally. Additionally, the patients fill in a questionnaire (SSQ12) to report perceived performance in their everyday life with their own devices. This is a post market study and all products used are CE marked and used in clinical practice worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adult BAHS users, minimum 18 years and maximum 75 years.
* Native English speakers.
* Patients that are already bilaterally implanted.
* Patients with a bilateral conductive or mixed conductive-sensorineural hearing loss.
* Experience with bilateral Ponto of at least 6 months.
* Patients that are using both their sound processors daily.
* PTA BC (at 0.5, 1, 2, 3 kHz) on both sides lower or equal to 65 dB HL.
* If the masked BC is available on the patient's journal, the average difference in masked BC (at 0.5, 1, 2, 4 kHz) between L and R ear should be lower than 15 dB.
* If the masked BC is not available on the patient's journal, the average difference in unmasked BC (at 0.5, 1, 2, 4 kHz) between L and R ear should be lower than 15 dB.

Exclusion Criteria:

* Not deemed suited by the principal investigator.
* If the physician assesses that the patient is not fit for trial participation at any stage.
* Audiogram at 1st visit shows too large masked BC thresholds (PTA BC - at 0.5, 1, 2, 3 kHz - on either side larger than 65 dB HL).
* Audiogram at 1st visit shows asymmetric masked BC thresholds (average difference in masked BC - at 0.5, 1, 2, 4 kHz - between L and R ear larger or equal to 15 dB).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Minimum Audible Angle test | 4 months
  Minimum angle at which noise bursts are accurately localized (Right/Left) in the unilateral and bilateral conditions

SECONDARY OUTCOMES:
SWIR test | 4 months
  Percentage of recalled words in the unilateral and bilateral conditions
SSQ12 | 4 months
  Subjective performance as measured by Speech, Spatial and Qualities of Hearing questionnaire (SSQ); 12 items with a scale from 0-10 where 0 represents "Not at all" and 10 represents "Perfect"

CONTACTS AND LOCATIONS:
Overall Officials: William Brassington, Principal Investigator — University Hospitals Birmingham, United Kingdom
Locations (1):
- Audiology Department, Nuffield House, University Hospitals Birmingham, Birmingham, West Midlands, United Kingdom